CLINICAL TRIAL: NCT04412174
Title: A Study of GC022F CAR-T Cell Immunotherapy for Relapsed or Refractory B- NHL
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: Gracell Biotechnology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGC011
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC022F (Experimental): The patients will receive GC022F CAR-T treatment. GC022F dosage ranges from 3×10^5 to 1×10^6 CAR+T/Kg.
  Interventions: Biological: GC022F

INTERVENTIONS:
Biological: GC022F — GC022F is a bispecific CAR-T cell immunotherapy that targeted CD19 and CD22. The dosage ranges from 3×10^5 to 1×10^6 CAR+T/Kg.

SUMMARY:
The study is an early, open, single-centered trial. The aim of this study is to evaluate the safety and tolerance of GC022F CAR-T cell immunotherapy in relapsed or refractory B-NHL. The investigators plan to include 18 subjects to receive GC022F therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Relapsed or refractory B cell non-Hodgkin's lymphoma (B-NHL): 1) Chemotherapy-refractory disease, defined as one or more of the following: a) No response to first-line therapy (primary refractory disease, subjects who are intolerant to first-line therapy chemotherapy are excluded): i. PD as the best response to first-line therapy; ii.SD as the best response after at least 4 cycles of first-line therapy (e.g., 4 cycles of R-CHOP) with SD duration no longer than 6 months from last dose of therapy; b) No response to second or greater lines of therapy: i. PD as the best response to most recent therapy regimen; ii. SD as the best response after at least 2 cycles of last line of therapy with SD duration no longer than 6 months from last dose of therapy; c) Refractory post-ASCT(autologous stem cell transplantation): i. Disease progression or relapsed ≤12 months of ASCT (must have biopsy proven recurrence in relapsed subjects); ii. If salvage therapy is given post-ASCT, the subject must have had no response to or relapsed after the last line of therapy; d) PD or SD as the best response after previous CAR-T therapy (at least 3 months ago); 2) Subjects must have received adequate prior therapy including at a minimum: anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20 negative, and an anthracycline containing chemotherapy regimen; for subjects with transformed FL must have received prior chemotherapy for follicular lymphoma and subsequently have chemotherapy-refractory disease after transformation to DLBCL; 3) At least 1 measurable lesion according to the Lugano Response Criteria (Cheson 2014). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy: a) For nodular lesions, longest diameter ≥15mm, no requirement for shortest diameter; b) For extranodal lesions (lesions other than lymph node and nodular lesions, including liver and spleen), longest diameter ≥10mm, no requirement for shortest diameter;
3. ECOG performance status ≤2 score;
4. Life expectancy≥12 weeks;
5. CD19 and/or CD22 positive expression demonstrated in tumor tissue;
6. Adequate organ function defined as: 1) Creatinine clearance (as estimated by Cockcroft Gault method)>60 mL/min; for male, creatinine clearance=[ (140-age)×weight(kg)]/[0.818×creatinine (μmol/L)] ; for female, creatinine clearance =[(140-age)×weight(kg)×0.85]/[0.818×creatinine (μmol/L)]; 2) Serum ALT/AST<2.5×ULN (for subjects with liver metastases, ALT/AST≤5×ULN); 3) Total bilirubin<1.5×ULN (for subjects with Gilbert's syndrome, total bilirubin≤ 3×ULN); 4) Left ventricular ejection fraction (LVEF)>50%, no evidence of clinically significant pericardial effusion as determined by an ECHO; 5) No clinically significant pleural effusion; 6) Baseline oxygen saturation >92% on room air;
7. Females of reproductive age must be in non-lactation period. Females of childbearing potential must have a negative hypersensitive serum pregnancy test. All subjects must use medical-approved-contraception (such as intrauterine device and contraceptive drugs) during the period of treatment and in 2 years after CAR-T infusion; males should avoid sperm donation;
8. Venous access can be established, peripheral blood mononuclear cells (PBMC) can be collected in researcher's judgement;
9. Agrees to sign informed consent form;
10. Be able to make good communication with researchers, willing and able to comply with the planned visit, complete the research according to regulations.

Exclusion Criteria:

1. Gastrointestinal involvement;
2. Active central nervous system (CNS) involvement;
3. Concomitant malignancy other than: cured non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, superficial bladder cancer, ductal carcinoma in situ, other malignancy whose disease-free survival exceeds 5 years;
4. Any result of the following virology tests is positive: HIV; HCV; HBsAg; or HBCAb positive with HBV DNA copies positive; TPPA;
5. Live vaccine ≤4 weeks prior to enrollment;
6. Autologous stem cell transplantation (ASCT) ≤6 weeks prior to enrollment, history of allogeneic hematopoietic stem cell transplantation (allo-HSCT);
7. Presence of complication that require systemic corticosteroids or other immunosuppressive drugs therapy during the trial in researcher's judgement;
8. CNS stereotactic radiotherapy ≤4 weeks prior to enrollment;
9. Toxicities related to previous therapy did not relieved to ≤1 grade, except hematological toxicity and alopecia;
10. Known life-threatening hypersensitivity to cyclophosphamide or fludarabine, or presence of other intolerant conditions, or severe allergic constitution;
11. Presence of active autoimmune disease (including but not limited to, systemic lupus erythematosus, sjogren syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, Hashimoto's thyroiditis, hypothyroidism which can be controlled by thyroid hormone replacement therapy is an exception);
12. Major surgical operation that require general anesthesia happened ≤4 weeks prior to enrollment, or did not be fully recovered and clinically stable prior to enrollment, or be anticipated to undergo major surgical operation that require general anesthesia during the study;
13. Usage of investigational drug ≤28 days prior to enrollment;
14. Any unstable cardiovascular disease happened ≤6 months prior to enrollment, including but not limited to, unstable angina, myocardial infarction, heart failure (NYHA grade ≥ III grade), severe arrhythmia that require drug interference, cardiac angioplasty/coronary stent implantation/cardiac bypass surgery ≤6 months prior to enrollment;
15. Presence of CNS disease or disease history, including epilepsy, cerebral Ischemia/bleeding, dementia, cerebellar disease, any autoimmune disease that involves CNS;
16. Any other condition that researcher think it is inappropriate for the subject to anticipate the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Type and incidence of DLT, incidence and severity of treatment related AE, CRS and Neurotoxicity (Safety and tolerability) | 2 years
  AE will be collected and graded according to ASTCT consensus(for Cytokine Release Syndrome, CRS and Immune Effector Cell-Associated Neurotoxicity Syndrome, ICANS) and CTCAE v5.0(for AE except CRS/ICANS)

SECONDARY OUTCOMES:
CAR copies of GC022F in peripheral blood, bone marrow, CSF and tumor tissue (amplification and persistence) | 2 years
  GC022F CAR copies in peripheral blood, tumor tissue, bone marrow and CSF will be measured by qPCR in 2 years.
CAR cells of GC022F in peripheral blood, bone marrow and CSF (amplification and persistence) | 2 years
  GC022F CAR cells in peripheral blood, bone marrow and CSF will be measured by FCM in 2 years.
Objective response rate (ORR) (efficacy) | 3 months
  ORR will be calculated as the percents of patients who achieved CR or PR.
Duration of Response (DOR) (efficacy) | 2 years
  DOR will be calculated as the time from the first assessment of CR or PR to the first assessment of relapse or death from any cause.
Progression-Free Survival (PFS) (efficacy) | 2 years
  PFS will be calculated as the time from CAR-T infusion to disease progression or death from any cause (whichever occurs first).
Overall Survival (OS) (efficacy) | 2 years
  OS will be calculated as the time from CAR-T infusion to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China